CLINICAL TRIAL: NCT05087641
Title: A Multicenter, Prospective Trial of the IAB in Adults Suffering From COPD/Emphysema
Acronym: IAB-1
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pulmair Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IAB1-CIP
Record Dates: First submitted 2021-09-28; First posted 2021-10-21 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Emphysema; Pulmonary Disease, Chronic Obstructive
Keywords: Bronchoscopic Lung Volume Reduction (BLVR)
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: This is an open-label (unblinded), multicenter, prospective trial of the Implantable Artificial Bronchus (IAB) in adults suffering from COPD/emphysema. There is no control group or comparator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- IAB System (Experimental): Patients will be treated with IAB(s)
  Interventions: Device: IAB System

INTERVENTIONS:
Device: IAB System — Bronchoscopic implantation of one or multiple IABs

SUMMARY:
The Pulmair Implantable Artificial Bronchus (IAB) is a device intended for implantation into the diseased bronchi of emphysema patients. The IAB is indicated for bronchoscopic treatment of adults with Chronic Obstructive Pulmonary Disease (COPD)/emphysema to relieve hyperinflation and allow bidirectional ventilation of the affected lobes.

The objective of this trial is to demonstrate a suitable benefit/risk profile to support a subsequent trial of the safety and effectiveness of the IAB to achieve its intended purpose.

The trial will enroll 24 subjects implanted with IAB(s), at no more than three study centers.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent
2. Diagnosis of COPD/emphysema
3. Age 40 to 75 years
4. Body Mass Index (BMI) less than 30 kg/m2
5. 6-minute walk Distance between 100 meters and 500 meters at baseline exam
6. Stable disease with less than 10 mg prednisone (or equivalent) daily
7. Non-smoking for 4 months prior to screening interview
8. FEV1 between 15% and 50% of predicted value at baseline exam
9. FEV1/Forced Vital Capacity (FVC) < 70%
10. RV > 175%
11. mMRC score ≥ 2

Exclusion Criteria:

1. Currently participating in another clinical study
2. Women of child-bearing potential
3. More than 2 COPD exacerbation episodes requiring hospitalization in the last year at screening
4. Any COPD exacerbations within 6 weeks of planned intervention
5. Two or more instances of pneumonia episodes in the last year at screening
6. Clinically significant mucus production or chronic bronchitis
7. Myocardial Infarction or unstable / uncontrolled congestive heart failure within 6 months of screening
8. Prior lung transplant, Lung Volume Reduction Surgery (LVRS), bullectomy or lobectomy
9. Clinically significant bronchiectasis
10. Unable to safely discontinue anti-coagulants or platelet activity inhibitors for 7 days
11. Uncontrolled pulmonary hypertension (systolic pulmonary arterial pressure > 45 mm Hg) or evidence or history of cor pulmonale as determined by recent echocardiogram (completed within the last 3 months prior to screening visit)
12. Suspected pulmonary nodule or lung cancer
13. High Resolution Computed Tomography (HRCT) collected per CT scanning protocol within the last 6 months of screening date and evaluated by clinical site personnel using 3D segmentation software shows:

    1. Large bullae encompassing greater than 30% of either lung
    2. Insufficient landmarks to evaluate the CT study using the software as it is intended
    3. All lobes are less than 25% parenchyma diseased (< -950 HU)
14. Any cardiac comorbidity which the PI believes would compromise the safety of the patient after an IAB implant
15. Total Lung Capacity (TLC) < 100% predicted at screening
16. Diffusing Capacity of Carbon Monoxide (DLCO) < 15% or > 50% of predicted value at screening
17. Partial pressure of carbon dioxide (PaCO2) > 50 mm Hg or Denver scale greater than 55 mm Hg on room air at screening
18. Partial pressure of oxygen (PaO2) < 45 mm Hg or Denver scale less than 30 mm Hg on room air at screening
19. Plasma cotinine level > 13.7 ng/ml or carboxyhemoglobin (arterial or ear lobe capillary) > 2.5% at screening
20. Any other conditions, which, in the opinion of the Investigator, would make the patient unsuitable for inclusion, or could interfere with the patient participating in or completing the study

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2024-03-27 (Actual); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Safety - Incidence of respiratory serious adverse events (SAEs) | From baseline to 90 days post implant (for endpoint evaluation)
  The primary endpoint is the occurrence of respiratory SAEs:
  * Acute asthma/bronchospasm requiring intensive/critical care unit admission
  * Acute COPD exacerbation (is acute onset, life-threatening, requires hospitalization)
  * Airway injury from IAB placement/migration/airway stenosis requiring surgical intervention
  * Death from procedure/IAB
  * Massive hemoptysis (est. >100 ml in 24hr requiring transfusion, surgery, or arterial embolization) from procedure/IAB
  * Pneumonia in treated lobe requiring hospitaliz., IV antibiotics, IAB removal
  * Pneumonia NOT in treated lobe (is life-threatening, acute onset, requires hospitaliz. & IV antibiotics)
  * Pneumothorax requiring surgery
  * Tension pneumothorax (is life-threatening, acute onset, requires hospitaliz. & treatment)
  * Respiratory failure requiring mechanical ventilatory support >24hr
  A thoracic SAE composite, based on number of subjects experiencing a thoracic SAE, will also be calculated and tabulated.

SECONDARY OUTCOMES:
Safety - Incidence of other serious adverse device effects (SADEs) | From baseline to 90 days post implant (for endpoint evaluation)
  All other SADEs are a secondary endpoint, made from the accumulation of adverse events (AEs) to be recorded as they occur regardless of the follow-up schedule.
Efficacy - Residual Volume (RV), absolute change | From baseline to 90 days post implant (for endpoint evaluation)
  Absolute change in Residual Volume (RV)
Efficacy - Residual Volume (RV), percent change | From baseline to 90 days post implant (for endpoint evaluation)
  Percent change in RV (% predicted)
Efficacy - Forced Expiratory Volume in one second (FEV1), absolute change | From baseline to 90 days post implant (for endpoint evaluation)
  Absolute change in FEV1
Efficacy - Forced Expiratory Volume in one second (FEV1), percentage change | From baseline to 90 days post implant (for endpoint evaluation)
  Percentage change in FEV1
Efficacy - Six-Minute Walk Distance (6MWD), absolute change | From baseline to 90 days post implant (for endpoint evaluation)
  Absolute change in 6MWD
Efficacy - Six-Minute Walk Distance (6MWD), percent change | From baseline to 90 days post implant (for endpoint evaluation)
  Percent change in 6MWD
Efficacy - Modified Medical Research Council (mMRC) dyspnea score, absolute change | From baseline to 90 days post implant (for endpoint evaluation)
  Absolute change in mMRC dyspnea score. Scores range from 0-4, with a decrease in score representing improved perception of disability attributable to dyspnea.
Efficacy - St. George's Respiratory Questionnaire (SGRQ) total score, absolute change | From baseline to 90 days post implant (for endpoint evaluation)
  Absolute change in SGRQ total score. Scores range from 0-100, with a decrease in score representing overall improvement in health, daily life, and perceived well-being.
Efficacy - St. George's Respiratory Questionnaire (SGRQ), percent change | From baseline to 90 days post implant (for endpoint evaluation)
  Percent change in SGRQ
Efficacy - COPD Assessment Test (CAT), absolute change | From baseline to 90 days post implant (for endpoint evaluation)
  Absolute changes in CAT. Scores range from 0-40, with a decrease in score representing decreased impact of cough, sputum, dyspnea, and chest tightness on overall health status.
Efficacy - COPD Assessment Test (CAT) Total Score, percent change | From baseline to 90 days post implant (for endpoint evaluation)
  Percent change in CAT Total Score
Efficacy - European Quality of Life, 5-Dimensional Test (EQ-5D) Summary Index, absolute change | From baseline to 90 days post implant (for endpoint evaluation)
  Absolute change in EQ-5D Summary Index. Index values range from 0-1, with a decrease in index value indicating an improvement in health-related quality of life.
Efficacy - European Quality of Life, 5-Dimensional Test (EQ-5D) Summary Index, percent change | From baseline to 90 days post implant (for endpoint evaluation)
  Percent change in EQ-5D Summary Index

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Goulart de Oliveira, MD, PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (3):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Brazil
- Thoraxklinik, University of Heidelberg, Heidelberg, Germany
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No